CLINICAL TRIAL: NCT01922895
Title: Novel Therapies in Moderately Severe Acute Alcoholic Hepatitis
Acronym: NTAH-Mod
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); The Cleveland Clinic (Other); University of Massachusetts, Worcester (Other); University of Louisville (Other)
Responsible Party: Principal Investigator, Mack Mitchell, Professor, Vice-Chair Internal Medicine, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: STU 092012-012; U01AA021893-01 (NIH)
Record Dates: First submitted 2013-08-12; First posted 2013-08-14 (Estimated); Results first posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Acute Alcoholic Hepatitis
Keywords: Alcoholic Hepatitis; MELD < 20; Probiotic; Nutritional Supplement; Lactobacillus Rhamnosus GG
MeSH Terms: conditions — Hepatitis, Alcoholic | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo for Probiotic (Placebo Comparator): Placebo capsule that matches the probiotic capsule in appearance will be given once daily for 180 days.
  Interventions: Drug: Placebo for Probiotic
- Lactobacillus Rhamnosus GG (Active Comparator): Dietary supplement capsule (Lactobacillus Rhamnosus GG) will be given once daily for 180 days.
  Interventions: Dietary Supplement: Lactobacillus Rhamnosus GG

INTERVENTIONS:
Dietary Supplement: Lactobacillus Rhamnosus GG — Probiotic nutritional supplement; Lactobacillus Rhamnosus GG
  Other Names: Culturelle
  Arms: Lactobacillus Rhamnosus GG
Drug: Placebo for Probiotic — Capsule manufactured without active ingredients.
  Other Names: Dummy capsule
  Arms: Placebo for Probiotic

SUMMARY:
This study is being done to find out whether a diet supplemented with a probiotic nutrient can improve alcoholic hepatitis and gut complications compared to routine standard care.

DETAILED DESCRIPTION:
Aim 1: Evaluate the effects of probiotic supplements on improvement in MELD score and gut mucosal integrity in patients with MELD < 21. Patients will be randomized to receive daily probiotics for 6 months and standard of care treatment or placebo with standard care.

Aim 2: Document the natural history of moderately severe alcoholic hepatitis. Patients who decline randomization will be offered the option of inclusion in the study prospectively for data collection purposes and research study procedures.

Aim 3: Create a data and tissue biorepository. This biorepository will serve as a national resource for studies related to acute alcoholic hepatitis.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide informed consent by subject or appropriate family member
2. Age between 21-70 years
3. Recent alcohol consumption > 50 g/d for > 6 months, continuing within two months before enrollment
4. At least 2 of the following symptoms or signs of acute alcoholic hepatitis: Anorexia, nausea, RUQ pain, jaundice, leukocytosis, hepatomegaly AND
5. Elevation of AST > 80 U/L, but < 500 U/L at the time of admission or within 3 days of baseline visit; AST > ALT and ALT < 200 U/L; total bilirubin > 3 mg/dL AND
6. Liver biopsy showing alcoholic hepatitis (steatohepatitis) OR ultrasound of liver showing increased echogenicity OR CT scan showing decreased attenuation of liver compared to spleen OR MRI showing fatty liver (decreased signaling intensity on T1 weighted images). If the liver biopsy (done within 60 days of inclusion) confirms diagnosis of AAH then inclusion e will be waived.
7. Model for End-Stage Liver Disease (MELD) <20
8. Willingness to utilize two reliable forms of contraception (both males and females of childbearing potential) from screening through the first six weeks of study.

Exclusion Criteria:

1. Hypotension with BP < 80/50 after volume repletion
2. Pregnancy; incarceration; inability to provide consent or lack of appropriate family member
3. Signs of systemic infection: Fever > 38o C and positive blood or ascites cultures on appropriate antibiotic therapy for > 3 days within 3 days of inclusion
4. Acute gastrointestinal bleeding requiring > 2 units blood transfusion within the previous 4 days
5. Undue risk from immunosuppression: Positive HBsAg; a positive skin PPD skin test or history of treatment for tuberculosis; history of any malignancy including hepatocellular carcinoma; known HIV infection
6. Treatment with corticosteroids or other immunosuppressive medications including specific anti-TNF therapy (not including pentoxifylline), calcineurin inhibitors for > 3 days within the previous 3 months.
7. Evidence of acute pancreatitis: CT evidence and/or amylase or lipase > 5 X upper limit of normal
8. Serious cardiac, respiratory or neurologic disease or evidence of autoimmune hepatitis, primary biliary cirrhosis, primary sclerosing cholangitis, Wilsons disease, hemochromatosis, secondary iron overload due to chronic hemolysis, alpha-1-antitrypsin deficiency
9. Acute or chronic kidney injury with serum creatinine > 3.0 mg/dl

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2013-08-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2021-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mack C Mitchell, M.D., Principal Investigator — U Texas Southwestern Medical Center
Locations (3):
- United States (3):
  - University of Louisville, Louisville, Kentucky
  - Cleveland Clinic, Cleveland, Ohio
  - U Texas Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vatsalya V, Feng W, Kong M, Hu H, Szabo G, McCullough A, Dasarathy S, Nagy LE, Radaeva S, Barton B, Mitchell M, McClain CJ. The Beneficial Effects of Lactobacillus GG Therapy on Liver and Drinking Assessments in Patients with Moderate Alcohol-Associated Hepatitis. Am J Gastroenterol. 2023 Aug 1;118(8):1457-1460. doi: 10.14309/ajg.0000000000002283. Epub 2023 Apr 11. PMID 37040544
- [Derived] Vatsalya V, Cave MC, Kong M, Gobejishvili L, Falkner KC, Craycroft J, Mitchell M, Szabo G, McCullough A, Dasarathy S, Radaeva S, Barton B, McClain CJ. Keratin 18 Is a Diagnostic and Prognostic Factor for Acute Alcoholic Hepatitis. Clin Gastroenterol Hepatol. 2020 Aug;18(9):2046-2054. doi: 10.1016/j.cgh.2019.11.050. Epub 2019 Dec 4. PMID 31811953

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lactobacillus Rhamnosus GG | Placebo for Probiotic
Started | 24 | 21
Completed | 18 | 7
Not Completed | 6 | 14
Not completed — Death | 0 | 1
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Lost to Follow-up | 5 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lactobacillus Rhamnosus GG | Placebo for Probiotic | Total
Number analyzed (Participants) | 24 | 21 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 21 | 45
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.2 (12.0) | 45.0 (9.4) | 44.6 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 20
  Male | 15 | 10 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 23 | 18 | 41
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 24 | 21 | 45

OUTCOME MEASURES:

1. Primary Outcome: MELD Score
Description: Change in MELD scoring system for assessing the severity of chronic liver disease; MELD (Model of End Stage Liver Disease) scoring system for assessing the severity of chronic liver disease; calculated from serum bilirubin, serum creatinine, and the international normalized ratio for prothrombin time (INR) MELD = 3.8[Ln serum bilirubin (mg/dL)] + 11.2[Ln INR] + 9.6[Ln serum creatinine (mg/dL)] + 6.4. MELD score range from 6-40 with higher scores indicating more severe liver disease and a worse outcome.
Time Frame: 30 days
Population: Four subjects from the LGG group and 8 subjects from the placebo group were lost to follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lactobacillus Rhamnosus GG | Placebo for Probiotic
Number analyzed (Participants) | 20 | 13
score on a scale | 14.25 (3.88) | 14.92 (6.08)

2. Secondary Outcome: MELD Score
Description: Change in MELD scoring system over 180 day study duration. MELD (Model of End Stage Liver Disease) scoring system for assessing the severity of chronic liver disease; calculated from serum bilirubin, serum creatinine, and the international normalized ratio for prothrombin time (INR) MELD = 3.8[Ln serum bilirubin (mg/dL)] + 11.2[Ln INR] + 9.6[Ln serum creatinine (mg/dL)] + 6.4. MELD score range from 6-40 with higher scores indicating more severe liver disease and a worse outcome.
Time Frame: 180 days
Population: 14 subjects from the LGG group and 17 subjects from the placebo group were lost to follow up by 180 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lactobacillus Rhamnosus GG | Placebo for Probiotic
Number analyzed (Participants) | 10 | 4
score on a scale | 11.0 (5.46) | 10.50 (3.11)

3. Secondary Outcome: MELD Score
Description: Change in MELD scoring system at 90 days study duration. MELD (Model of End Stage Liver Disease) scoring system for assessing the severity of chronic liver disease; calculated from serum bilirubin, serum creatinine, and the international normalized ratio for prothrombin time (INR) MELD = 3.8[Ln serum bilirubin (mg/dL)] + 11.2[Ln INR] + 9.6[Ln serum creatinine (mg/dL)] + 6.4. MELD score range from 6-40 with higher scores indicating more severe liver disease and a worse outcome.
Time Frame: 90 days
Population: 11 subjects from the LGG group and 16 subjects from the placebo group were lost to follow up by 90 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lactobacillus Rhamnosus GG | Placebo for Probiotic
Number analyzed (Participants) | 13 | 5
score on a scale | 11.62 (8.41) | 10.20 (3.89)

ADVERSE EVENTS:
Time Frame: 180 days
Arm/Group | Lactobacillus Rhamnosus GG | Placebo for Probiotic
All-Cause Mortality (participants affected / at risk) | 0/24 | 1/21
Serious Adverse Events (participants affected / at risk) | 17/24 | 15/21
Other Adverse Events (participants affected / at risk) | 16/24 | 15/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lactobacillus Rhamnosus GG (N=24) | Placebo for Probiotic (N=21)
Ascites (Cardiac disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Hepatitis alcoholic (Hepatobiliary disorders) | 1 | 0
Peritonitis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 2 | 0
Alcohol intolerance (Metabolism and nutrition disorders) | 0 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 2
Acute kidney injury (Renal and urinary disorders) | 9 | 2
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia bacterial (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rectal haemorrhage (Vascular disorders) | 0 | 1
Vaginal haemorrhage (Vascular disorders) | 1 | 0
Multiple conditions defined for single event (General disorders) | 0 | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lactobacillus Rhamnosus GG (N=24) | Placebo for Probiotic (N=21)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Ascites (Cardiac disorders) | 0 | 3
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 3
Pancreatitis (Gastrointestinal disorders) | 2 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 3 | 0
Lipase increased (Investigations) | 1 | 0
Alcohol intolerance (Metabolism and nutrition disorders) | 0 | 3
Anxiety (Psychiatric disorders) | 1 | 0
Drug dependence (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Urinary tract infection (Renal and urinary disorders) | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung infection (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Skin infection (Skin and subcutaneous tissue disorders) | 1 | 0
Multiple conditions defined for single event (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-11-16): https://cdn.clinicaltrials.gov/large-docs/95/NCT01922895/Prot_SAP_000.pdf
  • Informed Consent Form (2017-09-13): https://cdn.clinicaltrials.gov/large-docs/95/NCT01922895/ICF_001.pdf